CLINICAL TRIAL: NCT06909981
Title: Community-Based Engagement to Improve Lung Cancer Screening and Outcomes
Brief Title: Community-Based Engagement to Improve Lung Cancer Screening and Outcomes: The "Our Lungs Our Health" Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rian M. Hasson, MD, MPH, FACS, Associate Surgeon, Vice Chair for Workforce Development & Engagement, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24-715
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer Screening
Keywords: Lung Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung Cancer Screening (Experimental): Participants will complete a baseline questionnaire and undergo a shared decision-making with the study team to determine whether they will receive lung cancer screening. If the participant and team member determine that lung cancer screening should be performed, they will undergo screening. Regardless of whether lung cancer screening is performed, participants will undergo a debriefing conversation. An acceptability survey will be given to participants who underwent lung cancer screening. Those who undergo lung cancer screening will also be video-recorded speaking to their future selves as encouragement to get annual lung cancer screening. Imaging results will be returned to the participant and their care team within two weeks after lung cancer screening. Semi-structured interviews will also be performed with participants who underwent lung cancer screening between four and eight weeks after lung cancer screening. Video footage will be returned to patients after 48 weeks.
  Interventions: Radiation: Low-Dose Computed Tomography Scan

INTERVENTIONS:
Radiation: Low-Dose Computed Tomography Scan — Imaging of chest to screen for lung cancer.
  Other Names: CT Scan; LDCT Scan; CAT Scan

SUMMARY:
The main goal of this pilot study is to understand the impact of a mobile lung cancer screening clinics in individuals from neighborhoods and communities with less access to resources in Boston, Massachusetts who are at high risk for lung cancer. A secondary goal of this pilot study is to understand how social determinants of health impact these neighborhoods and communities. Another secondary goal of this pilot study is to see if video recording of participants speaking to their future selves and sending the videos back to participants to encourage them to get lung cancer screening after one year can be administered in a mobile lung cancer screening setting. The questions this study aims to answer are:

* Is mobile lung cancer screening is feasible and acceptable?
* Is collecting social needs data during the mobile lung cancer screening clinics feasible?
* Is creating video recordings of patients encouraging their future selves to get lung cancer screening after one year feasible?

Participants will:

* Complete an intake survey, providing information about their demographic, medical, and social needs information.
* Undergo a shared decision-making conversation to determine whether lung cancer screening should be done.
* Undergo lung cancer screening.
* Undergo a debriefing conversation and fill out an acceptability survey.
* Record a video speaking to their future selves about the importance of annual lung cancer screening, with the video to be sent back to them after roughly one year.
* Undergo a semi-structured phone interview between four and eight weeks after lung cancer screening date.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document prior to any study-related procedures.
* Willing to undergo treatment.
* Adults between the ages of 50 and 80 years.
* No recent CT imaging within the last year.
* Currently smokes tobacco or has quit smoking tobacco within the past 15 years.
* Has a tobacco smoking history of at least 20 pack years (i.e. one pack per day for the last 20 years or equivalent).
* Has never been diagnosed with lung cancer.

Exclusion Criteria:

* Adults/children less than 50 years, or greater than 80 years of age.
* Has never smoked tobacco.
* Has smoked tobacco but quit more than 15 years ago.
* Has a tobacco smoking history of less than 20 pack years.
* Presence of major comorbidity(ies) that could prevent treatment.
* Previous diagnosis of lung cancer.
* In the opinion of the investigator, the subject is not an appropriate candidate for the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of mobile lung cancer screening in target communities in Boston, Massachusetts. | During the intervention.
  This outcome will be assessed by calculating the raw count of individuals screened at each mobile clinic and the number of individuals unable to be screened due to time constraints.
Acceptability of mobile lung cancer screening in target communities in Boston, Massachusetts. | Between four and eight weeks after the intervention
  Acceptability will be assessed using semi-structured phone interviews with participants. Responses to questions, themes, and keywords will be analyzed to report attitudes regarding the intervention.

SECONDARY OUTCOMES:
Feasibility of collecting social determinants of health data during mobile lung cancer screening clinics in underserved communities in Boston, Massachusetts. | Pre-intervention
  Feasibility will be measured using the raw count of completed intake surveys.
Feasibility of administering a video-based intervention to encourage annual lung cancer screening | From enrollment until the end of the study.
  Participants who undergo mobile lung cancer screening will be recorded speaking to their future selves about the importance of annual lung cancer screening. The video footage will be returned to participants 48 weeks after mobile lung cancer screening to encourage the patient to schedule their next screening.